CLINICAL TRIAL: NCT04677257
Title: Coronary Physiology Testing in Acute Coronary Syndromes
Acronym: CoPhyTea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Prof. Paolo G Camici MD FACC, Prof Paolo G. Camici MD, FACC, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CoPhyTeA Trial
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: coronary microcirculation; coronary physiology; CMR
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: interventional, prospective, multicentre study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STEMI acute myocardial infarction treated with effective primary PCI (Experimental): STEMI patients treated with effective primary PCI to assess the ability of coronary physiology parameters (CFR and IMR) measured soon after recanalization to predict myocardial tissue characterization assessed with cardiac magnetic resonance (CMR) within a week of the acute event.
  Interventions: Procedure: PCI, invasive coronary physiology and CMR

INTERVENTIONS:
Procedure: PCI, invasive coronary physiology and CMR — Patients with acute STEMI will undergo invasive assessment of coronary physiology (IMR and CFR) following successful primary PCI and CMR within a week of the acute event

SUMMARY:
This is an interventional, prospective, multicenter study (5 IRCCS hospitals belonging to the Italian Cardiology Network) in patients with STEMI treated with successful primary PCI to assess the ability of coronary physiology parameters measured soon after recanalization to predict myocardial tissue characterization assessed with cardiac magnetic resonance (CMR) within a week of the acute event. Furthermore, patients will be followed up for a period of 12 months to assess the incidence of major adverse cardiovascular events (death, death from cardiovascular causes, re-infarction, new coronary revascularization interventions, development of heart failure) based on their stratification according to coronary physiology parameters.

DETAILED DESCRIPTION:
In the present study the investigators will enroll consecutive patients with STEMI acute myocardial infarction treated with successful primary PCI, to assess the ability of coronary physiology parameters, i.e. coronary flow reserve (CFR) and index of microvascular resistance (IMR) measured after recanalization to predict myocardial tissue characterization (MVO, MSI, IS, T2-rt, T1-rt and ECV) assessed with contrast CMR within a week of the acute event. Furthermore, the relationship between left ventricular end-diastolic pressure and of coronary physiology parameters will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with STEMI (defined according to ESC Guidelines 2017), with symptom onset within 12 hours (Class I), or between 12 and 48 hours (Class IIa), (1) successfully treated with primary PCI. (1)

Exclusion Criteria:

1. Patients with previous myocardial infarction in the territory of the infarct-related artery;
2. Patients with previous coronary artery bypass grafting;
3. Patients with cardiogenic shock at presentation;
4. Patients with need for mechanical support of the circulation;
5. Patients with known severe aortic stenosis / insufficiency;
6. Patients with known cardiomyopathy;
7. Patients with malignant neoplasm or systemic pathology with a "quoad vitam" prognosis of less than 1 year;
8. Patients affected by known active infectious diseases;
9. Women who are pregnant or breastfeeding;
10. Patients who are unable to express valid informed consent upon enrollment;
11. Patients with hypersensitivity to the active ingredients used for the study of coronary physiology (nitrates and adenosine);
12. Patients with specific contraindications to cardiac magnetic resonance imaging, including:

    * Patients with allergies and / or with other specific contraindications to the use of paramagnetic contrast media (gadolinium), including chronic renal failure with glomerular filtrate (eGFR) <30 mL / min;
    * Patients with non-resonance-compatible devices or who have undergone previous surgical interventions with placement of non-resonance-compatible vascular clips;
    * Claustrophobic patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Defining the predictive value of the classification of patients based on coronary physiology | 5 ± 2 days of the acute event.
  Establish the predictive value of the classification of patients based on coronary physiology measured in acute after primary PCI in patients with STEMI, on the incidence of microvascular obstruction (MVO) measured with CMR with contrast medium within 5 ± 2 days of the acute event.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo G Camici, MD, FACC, Principal Investigator — Ospedale San Raffaele
Locations (5):
- Italy (5):
  - IRCCS AOU San Martino, Genova
  - IRCCS Ospedale San Raffaele, Milan
  - IRCCS Centro Cardiologico Monzino, Milan
  - IRCCS Policlinico Gemelli, Roma
  - IRCCS Multimedica, Sesto San Giovanni

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benenati S, Montorfano M, Pica S, Crimi G, Ancona M, Montone RA, Rinaldi R, Gramegna M, Esposito A, Palmisano A, Tavano D, Monizzi G, Bartorelli A, Porto I, Ambrosio G, Camici PG. Coronary physiology thresholds associated with microvascular obstruction in myocardial infarction. Heart. 2024 Jan 29;110(4):271-280. doi: 10.1136/heartjnl-2023-323169. PMID 37879880